CLINICAL TRIAL: NCT06522594
Title: Randomized Embedded Multifactorial Adaptive Platform in ExtraCorporeal Membrane Oxygenation - Beta Receptor Modulation Trial
Brief Title: REMAP ECMO - Beta Receptor Modulation Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Christiaan Meuwese, Cardiologist-Intensivist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUCT 2024-511805-42
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Cardiogenic Shock
Keywords: Veno-Arterial ExtraCorporeal Membrane Oxygenation; Betablocker; Esmolol; Cardiogenic shock
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta receptor inhibition arm (Experimental): In the "beta receptor (BR) inhibition arm", patients are randomized to a biphasic strategy where BR stimulation is phased out and esmolol (BR blockade) is initiated in a sequential way. During a first phase, milrinone (a phosphodiesterase inhibitor which is routinely used in V-A ECMO supported patients) infusion will be initiated (if not already being given) at 0.25 mcg/kg/min and dobutamine dosages will be decreased every hour and eventually stopped according to the following sequence; 6 - 4 - 2 - 1 - 0 mcg/kg/min.
  In a second phase, esmolol is initiated with a dosage of 25 mcg/kg/min. The dose of the BB will be increased with increments of 25 mcg/kg/min every hour until reaching a heart rate between 50 and 70 bpm or a maximum dose of 200 mcg/kg/min. Prior to each dosage escalation, a reassessment of the hemodynamic situation will be done.
  The BR inhibition strategy will be continued until 48 hours after randomization or earlier when deemed necessary by the treating physician.
  Interventions: Drug: Esmolol
- Routine care arm (No Intervention): The dosage of dobutamine infusion is at the discretion of the treating physician but is typically continued until 48 hours after randomization. All other medication will be managed according to the needs of the patient at the discretion of the treating physician.

INTERVENTIONS:
Drug: Esmolol — A vey cardioselective, short-acting betablocker, with an ultra-short half life time.
  Arms: Beta receptor inhibition arm

SUMMARY:
In this phase 2, single center, randomized clinical pilot trial, investigators will study the effect of a strategy involving a reduction of beta receptor (BR) stimulation (by decreasing dobutamine dosages) and subsequent BR inhibition (through ultra-short acting betablockers), versus a (routine) strategy with continued BR stimulation through dobutamine infusion, on heart rate in patients with cardiogenic shock due to left- or bi-ventricular failure being supported by V-A ECMO.

DETAILED DESCRIPTION:
Despite the great benefits of Venoarterial ExtraCorporeal Membrane Oxygenation (V-A ECMO) and its rapidly increasing usage, even today, 30 till 70 percent of patients cannot be weaned from ECMO support and up to 50 percent of patients will eventually die in the first year. These high incidences of mortality and failure to wean from V-A ECMO support seem largely attributable to failure of the heart to recover in the context of inotropic drug administration and high sympathetic drive due to severe illness (further stressing an already failing heart). As V-A ECMO support creates a "safety window" where organ perfusion no longer relies on native cardiac output, therapeutic focus could be shifted to cardioprotective treatments. Cardioprotective treatments typically include beta blockers (BB) which have unequivocally shown benefits on mortality and morbidity in other patient categories with heart failure with reduced ejection fraction (HFrEF).

The investigators hypothesize that, in selected patients with cardiogenic shock undergoing V-A ECMO support, application of BBs is feasible and safe, and can effectively reduce heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Having received V-A ECMO support for severe circulatory insufficiency due to left- or bi-ventricular failure.
* ≤ 16 hours after initiation of V-A ECMO support
* Receiving ≥ 2 mcg/kg/min of dobutamine.
* Norepinephrine infusion ≤ 0.4 mcg/kg/min
* Heart rate ≥ 80 bpm (being sinus rhythm, atrial fibrillation or atrial flutter) after V-A ECMO initiation

Exclusion Criteria:

* Objection during the deferred consent procedure
* V-A ECMO usage confined to the period during surgery or another intervention (the ECMO was removed at the end of the intervention).
* Concomitant durable Left Ventricular Assist Device (LVAD)
* Polymorphic ventricular tachycardia necessitating BB therapy
* Isolated right ventricular failure (e.g. due to pulmonary embolism)
* Need of high dose dobutamine > 6.0 mcg/kg/min
* Epinephrine infusion
* Signs of insufficient trans cardiac flow:

  * Absence of aortic valve opening
  * Pulse pressure <10 mmHg (with intra-aortic balloon pump (IABP) standby)
  * Spontaneous contrast in the heart at echocardiography
* Contraindications for-, intolerance to- or allergy to esmolol
* Second- or third- degree AV block
* Pregnancy
* Life expectancy of less than 24 hours
* Participation in another randomized clinical trial (e.g. On Scene trial or Left Ventricular unloading trial)
* Inability to start study treatment within 4 hours after randomization
* Post heart transplantation patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Change (delta) in heart rate 24 hours after randomization. | 24 hours after randomization
  The average heart rate on basis of all observations during 5 minutes at both time points (t=0 and t=24h).

SECONDARY OUTCOMES:
Percentage of patients having received esmolol | after 48 hours
Vasopressor score | at baseline, 24 and 48 hours
  using the calculation as described in literature, excluding inotropic medication
Occurrence of new onset ventricular and/or atrial arrhythmias after randomization | during the first 48 hours
Left ventricular outflow tract velocity time integral (LVOT VTI) | at baseline, 24 and 48 hours
  Echocardiography parameters
Cardiac output | at baseline, 24 and 48 hours
  Pulmonary arterial catheter parameter
Stroke volume index | at baseline, 24 and 48 hours
  Pulmonary arterial catheter parameter
Pulmonary capillary wedge pressure | at baseline, 24 and 48 hours
  Pulmonary arterial catheter parameter
Central venous pressure | at baseline, 24 and 48 hours
  Pulmonary arterial catheter parameter
Mixed venous oxygen saturation (SvO2) | at baseline, 24 and 48 hours
  Pulmonary arterial catheter parameter
Lactate level | at baseline, 24 and 48 hours
Troponin | At 24 and 48 hours after randomization
  measured at baseline, 24- and 48- hours after randomization, and Area Under the Curve (AUC)
Myocardial oxygen consumption | At 24 and 48 hours after randomization
  Estimated by calculating the pressure volume (PV) area on basis of non-invasive PV loop assessments using echocardiography and pulmonary artery catheter measurements
Plasma NT-proBNP levels | At baseline and 48 hours after randomization
  Biomarker for cardiac stretch
Plasma Creatine Kinase MB levels | At baseline and 48 hours after randomization
  Biomarker for cardiac injury
FiO2 suppletion | At 24 and 48 hours after randomization
Plasma metanephrine levels | At baseline and 24 after randomization
Plasma normetanephrines levels | At baseline and 24 after randomization
Maximum median dosages of esmolol | after 48 hours
Ejection fraction (EF) | at baseline, 24 and 48 hours
  Echocardiography parameters
Tricuspid annular plane systolic excursion (TAPSE). | at baseline, 24 and 48 hours
  Echocardiography parameters
Positive End Expiratory Pressure (PEEP) level | At 24 and 48 hours after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan L. Meuwese, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Meuwese CL, Hermens JA, de Haan M, Braithwaite SA, Ramjankhan F, Buijsrogge MP, de Jonge N, Kirkels JH, de Jong M, Pasma W, Vromen-Wijsman JLP, Kraaijeveld AO, de Waal EE, Torn E, Platenkamp M, van der Heijden JJ, Cremer OL, van Dijk D, Donker DW. Twelve years of circulatory extracorporeal life support at the University Medical Centre Utrecht. Neth Heart J. 2021 Jul;29(7-8):394-401. doi: 10.1007/s12471-021-01552-z. Epub 2021 Mar 6. PMID 33675521
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Flather MD, Gollop ND. Understanding Mechanisms of Action of Beta-Blockers in Heart Failure With Reduced and Preserved Ejection Fraction. JACC Heart Fail. 2016 Feb;4(2):150-151. doi: 10.1016/j.jchf.2015.12.009. No abstract available. PMID 26823116
- [Background] Rahhal A, Omar AS, Aljundi A, Kasem M, Mahfouz A, Alyafei S. Successful Use of Intravenous B-blocker Therapy in Cardiogenic Shock Supported With Venoarterial Extracorporeal Membrane Oxygenation: A Case Series. Curr Probl Cardiol. 2022 Nov;47(11):101071. doi: 10.1016/j.cpcardiol.2021.101071. Epub 2021 Nov 26. PMID 34838902
- [Background] Brugts JJ, Manintveld O, Constantinescu A, Donker DW, van Thiel RJ, Nieman K, Jewbali LS, Zijlstra F, Caliskan K. Preventing LVAD implantation by early short-term mechanical support and prolonged inodilator therapy : A case series with acute refractory cardiogenic shock treated with veno-arterial extracorporeal membrane oxygenation and optimised medical strategy. Neth Heart J. 2014 Apr;22(4):176-81. doi: 10.1007/s12471-013-0509-5. PMID 24424723